CLINICAL TRIAL: NCT06184581
Title: Lithium Versus Lamotrigine in Bipolar Disorder, Type II - a Single Blinded Randomized Controlled Trial (the LiLa-Bipolar RCT)
Brief Title: Lithium Versus Lamotrigine in Bipolar Disorder, Type II
Acronym: LiLa-Bipolar
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Mental Health Centre Copenhagen, Bispebjerg and Frederiksberg Hospital (Other)
Responsible Party: Principal Investigator, Lars Vedel Kessing, professor, MD, DMSc., Mental Health Centre Copenhagen, Bispebjerg and Frederiksberg Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023-509607-32-00; 10.46540/2096-00007B (Other Grant/Funding Number: Independent Research Fund Denmark)
Record Dates: First submitted 2023-12-14; First posted 2023-12-28 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Bipolar II Disorder
MeSH Terms: conditions — Bipolar Disorder | interventions — Lithium Carbonate; lithium citrate; Lamotrigine

STUDY DESIGN:
Intervention Model Description: single-blinded two-armed, parallel randomized trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lithium (Experimental): tablet
  Interventions: Drug: Lithium Carbonate
- Lamotrigine (Active Comparator): tablet
  Interventions: Drug: Lamotrigine

INTERVENTIONS:
Drug: Lithium Carbonate — The trial is designed as a single-blinded two-armed, parallel randomized trial with randomization 1:1 to lamotrigine versus lithium.
  Other Names: lithium citrate
  Arms: Lithium
Drug: Lamotrigine — The trial is designed as a single-blinded two-armed, parallel randomized trial with randomization 1:1 to lamotrigine versus lithium.
  Arms: Lamotrigine

SUMMARY:
The investigators want in a 6-month randomized controlled trial (RCT) to compare effects of lithium versus lamotrigine on mood stabilization and other critical patient outcomes in patients with BDII.

DETAILED DESCRIPTION:
Although BDII is more prevalent and with a higher disease burden, including more and longer depressive episodes and lower functioning, than bipolar disorder, type I (BDI), effects of pharmacological treatment including the most frequently used drugs in clinical practice lithium and lamotrigine, is substantially understudied. The investigators want in a 6-month randomized controlled trial (RCT) to compare effects of lithium versus lamotrigine on mood stabilization and other critical patient outcomes in patients with BDII.

ELIGIBILITY:
Inclusion Criteria:

* Bipolar disorder, type II with diagnosis confirmed by SCAN interview
* Age 18-70 years
* Habile (i.e., able to give informed consent)

Exclusion Criteria:

* Past non-response or intolerance to lamotrigine or lithium with > 6 weeks treatment at an adequate dosage
* Currently taking mood stabilizers at enrollment in CADIC
* Severe chronic kidney disease
* Severe cardiac insufficiency
* Brugadas syndrome
* Severe hypothyroidism despite treatment
* Women who are pregnant, breastfeeding or planning pregnancy in near future.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-05-08 (Actual); Primary Completion 2027-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Mood stabilization | 6 (possibility of 12) months follow-up
  Mood Stabilization will be measured by a mood instability score reflecting the daily variability in self-monitored mood collected via the Monsenso app. Patients score their daily mood on a 9-point scale (-3 to +3); scores between -0.5 to 0.5 reflect normal variations, whereas scores of +1, +2 or +3 correspond to mildly, moderately, and severely increased mood and scores of -1, -2 or -3 correspond to mildly, moderately, and severely decreased mood. According to our established methodology, for each participant, we will estimate a mood instability score. Estimates of instability will be based on reading obtained via the Monsenso system which will prompt patients to complete daily mood ratings.

SECONDARY OUTCOMES:
Non-response | 6 (possibility of 12) months follow-up
  Add-on of Quetiapin >100mg/day or another antipsychotic drug, antidepressant drug, or inverse drug during the RCT-period or change from the allocated drug to lithium or lamotrigine
Depression | 6 months
  Clinically rated observer-based difference in depression scores over the six-month trial period on the Hamilton Depression Scale-6 items

CONTACTS AND LOCATIONS:
Locations (1):
- Psychiatric Center Copenhagen, Copenhagen, Denmark